CLINICAL TRIAL: NCT01531985
Title: Urine and Serum Biomarkers for Early Detection of Acute Kidney Injury Following Cardiopulmonary Bypass Surgery for Congenital Heart Disease in Children and Adults: A Pilot Study
Brief Title: Urine and Serum Biomarkers for Early Detection of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Earing, Associate Professor, Pediatrics, Cardiology, Medical College of Wisconsin
Other Study IDs: CHW 10/51; GC 1069
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Acute Kidney Injury; Cardiopulmonary Bypass; Biomarkers
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will be collected after the operation at 6 hours, 12 hours, 24 hours and 72 hours. The urine samples will be collected from your/your child's urinary catheter if one is in place for your/your child's regular hospital care, or by urine collected in a cup if you/your child do not have a urinary catheter. This study requires one blood samples of about 1 teaspoon, before surgery. The blood sample will be collected when other blood samples are drawn, to avoid extra needle sticks for blood. The extra blood collected, totaling about 1 teaspoon, is a safe amount for children over 2 years old.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out whether a combination of new urine tests and blood tests can show kidney injury in its early stages, before kidney failure sets in. If the investigators find new tests that show kidney injury in early stages, the investigators hope to start treating people with kidney injury earlier, to prevent kidney failure. You/your child are at higher risk for kidney injury and kidney failure than most other people, because of having operations with cardiopulmonary bypass (a machine that pumps your/your child's blood during the operation). This research is being done because there are no tests yet proven to show kidney injury before it leads to kidney failure.

The urine and blood tests the investigators are studying have each been shown to indicate some degree of kidney injury in certain people, but not with the accuracy needed to diagnose disease. The investigators think that the combination of urine and blood tests being tried in this research study may provide enough information to better diagnose kidney injury at an earlier stage.

About 20 persons over 2 years old up to adults will take part in this study. All will be from the Herma Heart Center of Children's Hospital of Wisconsin.

DETAILED DESCRIPTION:
Purpose: This will assess whether sensitive tests for urine or serum biomarkers are able to detect acute kidney injury following cardiopulmonary bypass surgery in the context of congenital heart disease.

Background: Acute kidney injury (AKI) is defined as an abrupt decrease in renal function resulting in retention of nitrogenous (urea and creatinine) and non-nitrogenous waste products. AKI is a common complication following cardiopulmonary bypass (CPB) surgery, occurring in up to 30% of adult patients following CPB surgery, increasing morbidity, mortality, and resource utilization.

Patients with cyanotic heart disease who undergo CPB surgery are also at risk of developing AKI. These patients require multiple surgeries over the course of their lifetime to correct their congenital cardiac lesions. Cyanosis alone causes a glomerulopathy characterized clinically by sub-nephrotic range proteinuria, with higher prevalence related to length of time prior to initial corrective procedures.

Pharmacological strategies for treatment of AKI have shown little efficacy in previous studies. Thus, recent studies have aimed to evaluate novel plasma and urinary biomarkers for early diagnosis of AKI, based on the hypothesis that outcomes may improve if AKI were identified and treatment initiated earlier. Urinary IL-18 and NGAL have been shown to be predictive markers of AKI after cardiopulmonary surgery in a pediatric population with a variety of congenital heart defects. This ultimately reduced detection time from 40 hours with conventional serum creatinine assays, to 4-6 hours with urinary IL-18 and NGAL. Serum Cystatin C has also been shown to be as reliable as serum creatinine in predicting kidney filtration levels, particularly for subjects with reduced muscle mass such as a population with congenital heart disease.

However, no study has evaluated the utility of such markers in a combined pediatric and adult congenital heart disease population. These patients are unique because of the multitude of CPB surgeries required throughout their lifetime, degree of life spent cyanotic and, thus, may differ in their susceptibility to cardiac surgery associated AKI.

Our long term goal is to evaluate the value of urinary and serum biomarkers for early detection of AKI in this unique patient population. Currently, the investigators propose to perform a pilot study to evaluate the feasibility of the study methods and to obtain preliminary data to assist in power calculations for a larger study.

Methods: The investigators will enroll a total of 20 patients undergoing pulmonary valve replacement. All patients will have a history of a conotruncal anomaly with previous corrective surgery requiring cardiopulmonary bypass. Enrollment will occur at the time of cardiology or cardiovascular surgery consultation.

After informed consent and assent is obtained, urine and serum samples will be collected for the study protocol. Urine specimens for creatinine, NGAL, and IL-18 will be collected pre-operatively for baseline measurement in addition to post-operatively at 6, 12, 24, and 72 hours. Cystatin C will be measured pre-operatively to assess chronic renal function. Serum creatinine will be measured pre-operatively and post-operatively at 12 hours and daily as part of usual clinical care.

Patients will be followed for 7 days after surgery or until the day of hospital discharge, whichever occurs first. Data collected from the hospital chart will include: demographics, medical and surgical history, type of surgical procedure, underlying congenital heart disease, baseline serum creatinine and renal function, serum creatinine(s) throughout hospitalization, daily urine output, need for dialysis, date of death or discharge. The primary endpoint is development of AKI based on serum creatinine reaching double baseline or requirement for acute dialysis, as described in the RIFLE- Risk, Injury, Failure, Loss, and End Stage Renal Disease- model of renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years of age or older
* Undergoing pulmonary valve replacement
* History of conotruncal anomaly ( including tetralogy of fallot, pulmonary atresia/VSD, truncus arteriosus, double outlet right ventricle)

Exclusion Criteria:

* unable to provide/obtain informed consent
* solid organ transplant recipients
* estimated baseline GFR < 30 ml/min (by MDRD-2)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will enroll a total of 20 patients undergoing pulmonary valve replacement with CPB. All patients will have a history of a conotruncal anomaly with previous corrective surgery requiring CPB.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Earing, MD, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin

REFERENCES:
- [Result] Buelow MW, Dall A, Regner K, Weinberg C, Bartz PJ, Sowinski J, Rudd N, Katzmark L, Tweddell JS, Earing MG. Urinary interleukin-18 and urinary neutrophil gelatinase-associated lipocalin predict acute kidney injury following pulmonary valve replacement prior to serum creatinine. Congenit Heart Dis. 2012 Sep-Oct;7(5):441-7. doi: 10.1111/j.1747-0803.2012.00662.x. Epub 2012 Apr 27. PMID 22537138